CLINICAL TRIAL: NCT02630212
Title: The Relationship Between ALDH2 and Aortic Dissection
Acronym: RALAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015QLMS37
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2018-12

CONDITIONS: Aortic Dissection
Keywords: Aortic dissection; Aldehyde dehydrogenase 2 polymorphism; Risk factor; aldehyde dehydrogenase 2
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 ml vein blood samples were collected from aortic dissection or controls in tubes containing EDTA. The samples would be centrifuged and saved in a -80℃ ultra-low temperature refrigerator.
  1 cm2 of aorta specimen were collected from patients operated on for Type A dissection, and refrigerated with liquid nitrogen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Chinese Han people undergoing coronary angiography in Qilu Hospital in corresponding period whose coronary arteries narrowing less than 50 percent.
- Aortic dissection: Chinese Han people diagnosed with aortic dissection in Qilu Hospital

SUMMARY:
The purpose of this study is to evaluate the impact of ALDH2 Glu504Lys polymorphism on aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Han people diagnosed with aortic dissection in Qilu Hospital

Exclusion Criteria:

* Aortic dissection based on trauma, connective tissue diseases and pregnancy
* Patients with tumor
* Patients with no written consensus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients diagnosed with aortic dissection in Qilu Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with different ALDH2 genotype | 1-30 days after samples collected
  DNA was extracted from venous blood;genomic DNA underwent PCR amplification; finally, PCR products were purified and directly sequenced by Invitrogen Corp or Biosune Corp.Then ALDH2 genotype was distinguished depend on a G-to-A missense mutation on exon 12 of ALDH2 gene.

SECONDARY OUTCOMES:
Concentration of inflammatory factors in blood and aortic specimen | 1-30 days after samples collected
  Concentration of 4-HNE、MMP-2、MMP-9 detected by elisa kit、IHC or western blot in relevant specimen.
ALDH2 activity | 1-30 days after samples collected
  Activity of ALDH2 was detected in blood and aortic specimen depend on its reducibility of NAD+

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China